CLINICAL TRIAL: NCT04445558
Title: Study of Two Modalities of Dialysis and Nutrition on the Nutritional Status of Malnourished Chronic End-stage Renal Disease Patients Dependent on Intradialytic Parenteral Nutrition
Brief Title: Study of 2 Modalities of Dialysis and Nutrition on the Nutritional Status of Malnourished Chronic Renal Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A01267-32
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Membrane PEPA® (Experimental): Patient will use the membrane PEPA® for the dialysis
  Interventions: Dietary Supplement: oral nutritional supplementation
- Standard membrane of dialysis (Active Comparator): Patient will use a standard membrane for the dialysis
  Interventions: Dietary Supplement: intradialytic parenteral nutrition

INTERVENTIONS:
Dietary Supplement: oral nutritional supplementation — Adjunction of oral nutritional supplementation
  Arms: Membrane PEPA®
Dietary Supplement: intradialytic parenteral nutrition — Adjunction of intradialytic parenteral nutrition
  Arms: Standard membrane of dialysis

SUMMARY:
Describe the impact of dialysis by high permeability and adsorbent membrane (PEPA®) associated with oral nutritional supplementation on the nutritional status of malnourished chronic end-stage renal disease patients dependent on intradialytic parenteral nutrition.

DETAILED DESCRIPTION:
The study proposes to compare the nutritional state after 6 months of dialysis with standard membrane associated with intradialytic parenteral nutrition (retrospective phase) with the nutritional state after 6 months of dialysis with high permeability membrane associated with oral nutritional supplementation (prospective phase).

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal failure, on hemodialysis for at least 12 months;
* Hemodialysis patient in 3 weekly sessions on a device with a standard permeability membrane (polysulfone, polyethersulfone or polyartylethersulfone type);
* Malnourished patient, on intradialytic parenteral nutrition for at least 6 months;
* Patient who may benefit, according to the doctor, from a change in dialysis and nutrition strategy:
* Patient who signed an informed consent form to participate in the study

Exclusion Criteria:

* Known allergy to PEPA® ;
* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision);
* Patient with a chronic infection in progress;
* Patient with life expectancy <6 months according to the investigator;
* Inability to understand information related to the study (linguistic, psychological, cognitive reason, etc.);
* Pregnant woman or likely to be (of childbearing age, without effective contraception) or breastfeeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Evolution of the nutritional status | Month 6
  The main endpoint is the evolution between M0 and M6 of the nutritional status measured by the serum albumin level.

SECONDARY OUTCOMES:
Evolution of nutritional assessment | Month 6
  Evolution of the percentage of weight loss (in Kg)
Appearance of adverse events | Month 6
  Incidence and characteristics of adverse events / effects
Measure of the Quality of life | Month 6
  Evolution of the quality of life, evaluated by the EORTC QLQ-C30 questionnaire of the quality of life with 28 questions with 4 possible answers from "not at all" to "a lot of"

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé La Louvière, Lille, France

IPD SHARING:
Plan to Share IPD: No